CLINICAL TRIAL: NCT04842539
Title: Single Session of Fecal Microbiota Transplantation in Decompensated Cirrhosis: An Open-label Randomized Control Trial
Brief Title: Fecal Microbiota Transplantation in Decompensated Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Radha K Dhiman, Professor of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT/IEC2018/2076
Record Dates: First submitted 2021-04-03; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Liver Cirrhosis
Keywords: End-stage liver disease; Stool therapy; Microbiota; Related stool donor; Prognostic scores; Complications; Ammonia; Cytokines; Outcomes
MeSH Terms: conditions — Liver Cirrhosis; End Stage Liver Disease | interventions — Fecal Microbiota Transplantation; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT Arm (Experimental): FMT Arm:30 grams stool homogenized with 100 mL normal saline and filtered administered a single time via nasojejunal tube.
  Interventions: Other: Fecal Microbiota Transplantation
- Standard of care (SOC) Arm (Other): Standard of care treatment with nutritional supplementation and other supportive care
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Fecal Microbiota Transplantation — In the Fecal Microbiota Transplantation procedure 100 ml volume of strained and filtered stool will be delivered through a nasojejunal tube.The recipient patient will be kept nil per oral for at least 4 hours prior to the stool instillation. 100 mL of freshly prepared stool suspension will be given.
  Arms: FMT Arm
Other: Standard of care — Nutritional supplementation and other supportive measures as per standard guidelines
  Arms: Standard of care (SOC) Arm

SUMMARY:
Cirrhosis of the liver is the culmination point of long-standing chronic liver disease hallmarked by the cardinal features of liver fibrosis and portal hypertension. The prognosis of patients with cirrhosis is punctuated by the onset of complications which denote the stage of decompensation characterized by ascites, hepatic encephalopathy (HE), and variceal bleeding.

Patients with cirrhosis have been demonstrated to have significant changes in their gut microbiota characterized by alteration in the intestinal microbiome (gut dysbiosis) as well as small intestinal bacterial overgrowth (SIBO). Gut dysbiosis has been closely linked to the complications associated with decompensated cirrhosis. Several studies have documented the alteration of gut microbiota in patients with hepatic encephalopathy.

Therapeutic modalities that restore normal gut flora and stabilize the gut liver axis are being extensively studied in the management of cirrhosis and its complications. Antibiotics, probiotics, and long-chain fatty acid supplementation are being evaluated as methods to restore the gut dysbiosis and consequently limit progressive liver damage.

Fecal Microbiota Transplantation (FMT) involves the infusion of intestinal microorganisms by the transfer of stool from a healthy individual into a diseased individual for restoration of normal intestinal flora.The ultimate goal of FMT is to replace aberrant native microbiota with a stable community of donor microorganisms. The treatment is based on the premise that an imbalance in the community of microorganisms residing in the gastrointestinal tract (i.e., dysbiosis) is associated with specific disease states. FMT has been well-established as a treatment modality to stably modify the gut microbiome and has been shown to be safe and efficacious in several disease states resulting from gut dysbiosis.

With this background, a trial is proposed to determine whether an FMT from a healthy donor to a patient with advanced cirrhosis improves overall survival and prognosis.

ELIGIBILITY:
Inclusion Criteria:

Age 18-65 years Decompensated cirrhosis (of any etiology) based on clinical, radiological, or histological criteria Model for end-stage liver disease (MELD scores) between 12-21 were included.

Exclusion Criteria:

Ongoing bacterial infection requiring antibiotics Antibiotics/pre-pro biotics within the last 14 days, t Significant alcohol intake in the previous two months, Recent (<14 days) history of spontaneous bacterial peritonitis, HE or variceal bleed, History of substance abuse or psychiatric illness, HIV infection, Pregnant patients, Hepatocellular carcinoma or other known malignancy, t Prior liver transplantation or bariatric surgery, Immunosuppression, Inflammatory bowel disease Celiac disease, History of allergy to food substances

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Survival | 180 day
  180 days

SECONDARY OUTCOMES:
Change in Child Turcotte Pugh Score | 180 days
Change in MELD score | 180 days
Change in MELD Na score | 180 days
Change in ammonia level | 28 days
Change in Interleukin level | 28 days
Number of patients with incident Hepatic encephalopathy | 180 days
Number of patients with incident Variceal Bleed | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT04842539/Prot_SAP_000.pdf